CLINICAL TRIAL: NCT06422299
Title: Developing and Testing an Online Intervention for Decreasing Alcohol and Cannabis Misuse and Increasing Healthy Relationship Skills Among Young Adult Couples: A Comprehensive Mixed-methods Approach
Brief Title: Developing and Testing an Online Intervention for Alcohol and Cannabis Misuse and Healthy Relationship Skills Among Young Adult Couples
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Katherine Walukevich-Dienst, Acting Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00017992; K23AA031034-01 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Drinking; Cannabis Use; Couples
Keywords: alcohol use, cannabis use, couples, healthy relationships, young adults
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online, couples-based intervention (Experimental): A novel, brief online intervention for young adults community couples who engage in alcohol and cannabis co-use.
  Interventions: Behavioral: Online, couples-based intervention
- Assessment-only control (No Intervention): Couples in the control condition will not receive an intervention.

INTERVENTIONS:
Behavioral: Online, couples-based intervention — During Phase 1 of the present study, the intervention will be iteratively developed using a rigorous, user-centered design approach through integration of knowledge gained from Phase 1 dyadic analyses and qualitative interviews, and existing gold-standard treatments for substance use among couples, including Integrative Behavioral Couples Therapy (IBCT; Christensen & Doss, 2016) and Behavioral Couples Therapy for Alcohol (ABCT; McCrady et al, 1995) and substance use brief interventions for young adults (Halladay, et al., 2019; Tanner-Smith et al., 2015).
  Arms: Online, couples-based intervention

SUMMARY:
The goal of this clinical trial is to develop and test a brief online intervention to reduce alcohol and cannabis misuse and improve healthy relationship skills among young adult couples. The main questions it aims to answer are:

* Will the intervention be feasible and acceptable to young adult couples?
* Will the intervention demonstrate initial efficacy in reducing risky substance use and increasing relationship functioning?

Eligible couples will complete a virtual baseline session and be randomized to intervention condition (online intervention with 3-5 weeks of self-paced modules) or control condition (no intervention). Couples will complete two follow-up surveys (post-assessment - approximately 5 weeks after baseline, 3-month). Couples in the control condition will be offered the intervention after 3-month follow-up.

Researchers will compare intervention and control groups to see if there there is a difference between the groups on substance misuse and relationship functioning at post-assessment and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Both partners in the couple are 18-29 years old
* In a committed romantic relationship (e.g., dating seriously, cohabiting, married) with each other for at least 3 months
* Face-to-face contact their partner at least 5 days per week
* Live in Washington State
* Have a valid email address and access to a cell phone
* Report alcohol and cannabis co-use at least three times in the past month
* Willingness to: complete online surveys during the allotted time frames, receive text messages and emails from the project, complete a baseline session, and participate during the same time period as their partner

Exclusion Criteria:

* Couples who endorse any perpetration or receipt of severe interpersonal aggression during screening will be excluded and provided with resources

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Heavy episodic and high intensity drinking | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Alcohol use - number of days in the past month participant engaged in heavy episodic drinking (4+/5+ drinks in one occasion for women/men) and high intensity drinking (8+/10+ drinks in one occasion for women/men)
Daily Drinking Questionnaire (DDQ) | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Alcohol use - Average total drinks per week will be calculated as the sum of the total number of drinks reported.
Daily Marijuana Questionnaire (DMQ) | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Cannabis use - Average total hours high from cannabis per week will be calculated as the sum of the total hours high reported
Intensity of Marijuana Use | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Cannabis use intensity - Average number of times used cannabis per day will be calculated as the mean number of times participant reports using cannabis per each day of a typical week in the past month
Perceived Program Effects on Healthy Relationship Self-Efficacy items | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Healthy relationship self-efficacy - 3 items assessing perceived intervention impacts on healthy relationship self-efficacy scored 0=strongly disagree to 5=strongly agree. Scores will be summed, total scores will range from 0 to 15, with higher scores indicating greater healthy relationship self-efficacy
Couples Satisfaction Index | Screening, baseline, approximately 5 weeks after baseline, 3-month followup
  Relationship satisfaction - sum of 4 items ranges from 0 to 21, higher scores indicate greater relationship satisfaction

REFERENCES:
- [Background] Patrick ME. A Call for Research on High-Intensity Alcohol Use. Alcohol Clin Exp Res. 2016 Feb;40(2):256-9. doi: 10.1111/acer.12945. No abstract available. PMID 26842244
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Lee CM, Kilmer JR, Neighbors C, Atkins DC, Zheng C, Walker DD, Larimer ME. Indicated prevention for college student marijuana use: a randomized controlled trial. J Consult Clin Psychol. 2013 Aug;81(4):702-9. doi: 10.1037/a0033285. Epub 2013 Jun 10. PMID 23750464
- [Background] Patrick ME, Veliz PT, Terry-McElrath YM. High-intensity and simultaneous alcohol and marijuana use among high school seniors in the United States. Subst Abus. 2017 Oct-Dec;38(4):498-503. doi: 10.1080/08897077.2017.1356421. Epub 2017 Jul 20. PMID 28726580
- [Background] Scott ME, Moore KA, Fish H, Benedetti A, Erikson S. OPRE Report #2015-65a. Prepared by Child Trends. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services. 2015. https://www.acf.hhs.gov/sites/default/files/documents/b_hmre_recommended_outcome_measures_for_adolescents_508_0.pdf
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329